CLINICAL TRIAL: NCT03706833
Title: Edwards PASCAL TrAnScatheter Valve RePair System Pivotal Clinical Trial (CLASP IID/IIF): A Prospective, Multicenter, Randomized, Controlled Pivotal Trial to Evaluate the Safety and Effectiveness of Transcatheter Mitral Valve Repair With the Edwards PASCAL Transcatheter Valve Repair System Compared to Abbott MitraClip in Patients With Mitral Regurgitation
Brief Title: Edwards PASCAL CLASP IID/IIF Pivotal Clinical Trial
Acronym: CLASP IID/IIF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-07
Record Dates: First submitted 2018-10-10; First posted 2018-10-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Mitral Valve Disease; Mitral Regurgitation; Mitral Insufficiency; Functional Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- Edwards PASCAL System - CLASP IID (Experimental): Transcatheter mitral valve repair with the Edwards PASCAL System in patients with degenerative mitral regurgitation
  Interventions: Device: Edwards PASCAL System
- Abbott Mitraclip System - CLASP IID (Active Comparator): Transcatheter mitral valve repair with the Abbott Mitraclip System in patients with degenerative mitral regurgitation
  Interventions: Device: Abbott Mitraclip System
- Edwards PASCAL System - CLASP IIF (Experimental): Transcatheter mitral valve repair with the Edwards PASCAL System in patients on guideline directed medical therapy with functional mitral regurgitation
  Interventions: Device: Edwards PASCAL System
- Abbott Mitraclip System - CLASP IIF (Active Comparator): Transcatheter mitral valve repair with the Abbott Mitraclip System in patients on guideline directed medical therapy with functional mitral regurgitation
  Interventions: Device: Abbott Mitraclip System
- Edwards PASCAL System - Single-Arm Registry (Experimental): Transcatheter mitral valve repair with the Edwards PASCAL System in patients with mitral regurgitation who were deemed non-randomizable by a central screening committee (CSC) due to complex anatomical features described in the current MitraClip Instructions for Use (IFU) but were considered suitable for the PASCAL system.
  Interventions: Device: Edwards PASCAL System

INTERVENTIONS:
Device: Edwards PASCAL System — Transcatheter mitral valve repair with the Edwards PASCAL System
  Other Names: Transcatheter Mitral Valve repair (TMVr)
  Arms: Edwards PASCAL System - CLASP IID; Edwards PASCAL System - CLASP IIF; Edwards PASCAL System - Single-Arm Registry
Device: Abbott Mitraclip System — Transcatheter mitral valve repair with the Abbott Mitraclip System
  Other Names: Transcatheter Mitral Valve repair (TMVr)
  Arms: Abbott Mitraclip System - CLASP IID; Abbott Mitraclip System - CLASP IIF

SUMMARY:
To establish the safety and effectiveness of the Edwards PASCAL Transcatheter Valve Repair System in patients with degenerative mitral regurgitation (DMR) who have been determined to be at prohibitive risk for mitral valve surgery by the Heart Team, and in patients with functional mitral regurgitation (FMR) on guideline directed medical therapy (GDMT)

DETAILED DESCRIPTION:
A prospective, multicenter, randomized, controlled pivotal trial to evaluate the safety and effectiveness of transcatheter mitral valve repair with the Edwards PASCAL Transcatheter Valve Repair System compared to Abbott MitraClip in patients with degenerative mitral regurgitation (DMR) who have been determined to be at prohibitive risk for mitral valve surgery by the Heart Team, and in patients with functional mitral regurgitation (FMR) on guideline directed medical therapy (GDMT)

Patients will be seen for follow-up visits at discharge, 30 days, 6 months, and annually through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen (18) years of age or older
* Patient is able and willing to give informed consent and follow protocol procedures, and comply with follow-up visit requirements.
* Patient is determined to be at prohibitive risk for mitral valve surgery by the heart team (CLASP IID cohort only).
* Patient is on stable heart failure medications/Guideline Directed Medical Therapy (CLASP IIF cohort only)
* Patient is determined to be a candidate for transcatheter mitral valve repair by the heart team for both PASCAL and MitraClip
* Mitral regurgitation (3+ to 4+) by echo
* Suitable valve and regurgitant jet morphology
* Elevated corrected BNP > 400 pg/ml or corrected NT-pro BNP of > 900 pg/ml or heart failure hospitalization within the past 12 months (CLASP IIF cohort only)
* LVEF ≥ 20% (and ≤ 50%; CLASP IIF cohort only)

Exclusion Criteria:

* Patient in whom a TEE is contraindicated or screening TEE is unsuccessful
* Mitral valve anatomy which may preclude proper PASCAL or MitraClip access, use and/or deployment or sufficient reduction in mitral regurgitation
* Patient with refractory heart failure requiring advanced intervention (i.e. left ventricular assist device, Status ≤5 heart transplantation) (ACC/AHA Stage D heart failure)
* Clinically significant, untreated coronary artery disease
* Recent stroke
* Other severe valve disorders requiring intervention
* Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months
* Any prior mitral valve surgery or transcatheter mitral valve procedure (excluding chordal replacement or surgical annuloplasty repair)
* Severe tricuspid regurgitation or tricuspid valve disease requiring surgery
* Active rheumatic heart disease or rheumatic etiology for MR
* Severe aortic stenosis or regurgitation
* Known history of untreated, severe carotid stenosis
* Recent deep vein thrombosis (DVT) or pulmonary embolism (PE)
* Severe COPD
* Pregnant or planning pregnancy within next 12 months. Note: Female patients of childbearing potential need to have a negative pregnancy test performed within 14 days prior to intervention and be adherent to an accepted method of contraception
* Concurrent medical condition with a life expectancy of less than 12 months in the judgment of the Investigator
* Patient is currently participating in another investigational biologic, drug or device clinical study where the primary study endpoint was not reached at time of enrollment
* Other medical, social, or psychological conditions that preclude appropriate consent and follow-up, including patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1247 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
PASCAL is not inferior to MitraClip with respect to the proportion of patients with major adverse events (MAE). The primary safety endpoint is a composite of Major Adverse Events (MAEs). | 30 days.
PASCAL is not inferior to Mitraclip with respect to the proportion of patients with MR severity reduction as measured by echocardiography using a scale of 0-4+ for the CLASP IID Cohort. | 6 months
PASCAL is not inferior to Mitraclip with respect to the time to first heart failure hospitalization or death for the CLASP IIF Cohort only. | From date of randomization until date of first heart failure hospitalization or death, through 5 year follow-up

SECONDARY OUTCOMES:
Rates of various adverse events | 6 months; 12 months
  Rates of various adverse events at 6 and 12 months
Functional Improvement (increase in 6 minute walk test in meters) | 30 days , 6 months, 1 year
  Increase in 6 minute walk test in meters
Functional improvement (quality of life) as assessed using the Kansas City Cardiomyopathy Questionnaire through 2 years | 30 days , 6 months, 1 year, 2 year
  Number of points of improvement on a scale of 0-100 in Kansas City Cardiomyopathy Questionnaire, with higher scores associated with higher Quality of Life
Functional improvement (quality of life) as assessed by number of points of improvement on the Short Form Health Survey (SF-36) questionnaire through 2 years | 30 days, 6 months, 1 year, 2 year
  Number of points of improvement on a scale of 0-100 in Short Form Health Survey (SF-36) questionnaire, with higher totals associated with higher Quality of Life
Functional improvement (quality of life) as assessed by number of points of improvement on the Short Form Health Survey (EQ-5D-5L) questionnaire through | 30 days, 6 months, 1 year, 2 year
  Number of points of improvement on a scale of 1-100 in Short Form Health Survey (EQ-5D-5L) questionnaire, with higher totals associated with higher Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lim, MD, Principal Investigator — University of Virginia; Robert Smith, MD, Principal Investigator — The Heart Hospital Baylor Plano; Linda Gillam, MD, Principal Investigator — Morristown Medical Center; Vinod Thourani, MD, Principal Investigator — Piedmont Healthcare; Paul Grayburn, MD, Principal Investigator — The Heart Hospital Baylor Plano; Brian K Whisenant, MD, Principal Investigator — Intermountain Medical Center; Jörg Hausleiter, MD, Principal Investigator — LMU München, Campus Gorsshadern; Ralph Stephan von Bardeleben, MD, Principal Investigator — / Universitätsmedizin Mainz- Zentrum für Kardiologie
Locations (87):
- United States (69):
  - Banner University Medical Center, Phoenix, Arizona
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - TMC Healthcare, Tucson, Arizona
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine, Orange, California
  - Sutter Medical Center-Sacramento, Sacramento, California
  - Sutter Bay Area, San Francisco, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - The Cardiac and Vascular Institute Research Foundation, Gainesville, Florida
  - Mount Sinai, Miami Beach, Florida
  - NCH Healthcare System Naples, Naples, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University Hospital and Emory University Hospital Midtown, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St. Vincent Heart Center, Carmel, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Woman's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - St.Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers-RWJMS, New Brunswick, New Jersey
  - Albany Medical College, Albany, New York
  - State University of New York at Buffalo, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Lenox Hill Hospital and North Shore University, New York, New York
  - Rochester General Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Cardiovascular, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania/Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Pinnacle Health Cardiovascular Institute/ UPMC Pinnacle Harrisburg, Wormleysburg, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - CVA Heart Institute Kingsport, Kingsport, Tennessee
  - Baptist Memorial Hospital Memphis, Memphis, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Saint Thomas Heart at Saint Thomas West, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (5):
  - St. Pauls Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ) ULaval, Québec
- Germany (12):
  - Klinik für Allgemeine und Interventionelle Kardiologie/Angiologie, Herz- und Diabeteszentrum NRW, Universitätsklinik der Ruhr-Universität Bochum, Bad Oeynhausen
  - Herzzentrum Universitätsklinikum Koln, Cologne
  - Herrzentrum Dresden GmbH Universitätklinik an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Essen (AöR) Klinik für Kardiologie und Angiologie am Westdeutschen Herz- und Gefäßzentrum, Essen
  - Universitätsklinikum Gießen Medizinische Klinik I, Innere Medizin/ Kardiologie, Giessen
  - Universitäres Herzzentrum Hamburg GmbH (UHZ) Klinik und Poliklinik für Allgemeneine und Interventionelle Kardiologie, Hamburg
  - Universitätsklinikum Heidelberg Klinik für Kardiologie, Angiologie, Pneumologie, Heidelberg
  - Herzzentrum Leipzig Universitätsklinik für Kardiologie, Leipzig
  - Zentrum für Kardiologie - Kardiologie I Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz
  - Medizinische Klinik I LMU München Campus Grosshadern, München
  - Helios Klinikum Siegburg, Siegburg
  - ULM University Zentrum für Innere Medizin Klinik für Innere Medizin II, Ulm
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcoff L, Koulogiannis K, Aldaia L, Mediratta A, Chadderdon SM, Makar MM, Ruf TF, Gossler T, Zaroff JG, Leung GK, Ku IA, Nabauer M, Grayburn PA, Wang Z, Hawthorne KM, Fowler DE, Dal-Bianco JP, Vannan MA, Bevilacqua C, Meineri M, Ender J, Forner AF, Puthumana JJ, Mansoor AH, Lloyd DJ, Voskanian SJ, Ghobrial A, Hahn RT, Mahmood F, Haeffele C, Ong G, Schneider LM, Wang DD, Sekaran NK, Koss E, Mehla P, Harb S, Miyasaka R, Ivannikova M, Stewart-Dehner T, Mitchel L, Raissi SR, Kalbacher D, Biswas S, Ho EC, Goldberg Y, Smith RL, Hausleiter J, Lim DS, Gillam LD; CLASP IID Pivotal Trial Investigators. Echocardiographic Outcomes With Transcatheter Edge-to-Edge Repair for Degenerative Mitral Regurgitation in Prohibitive Surgical Risk Patients. JACC Cardiovasc Imaging. 2024 May;17(5):471-485. doi: 10.1016/j.jcmg.2023.09.015. Epub 2023 Dec 13. PMID 38099912
- [Derived] Hausleiter J, Lim DS, Gillam LD, Zahr F, Chadderdon S, Rassi AN, Makkar R, Goldman S, Rudolph V, Hermiller J, Kipperman RM, Dhoble A, Smalling R, Latib A, Kodali SK, Lazkani M, Choo J, Lurz P, O'Neill WW, Laham R, Rodes-Cabau J, Kar S, Schofer N, Whisenant B, Inglessis-Azuaje I, Baldus S, Kapadia S, Koulogiannis K, Marcoff L, Smith RL; PASCAL IID Registry Investigators. Transcatheter Edge-to-Edge Repair in Patients With Anatomically Complex Degenerative Mitral Regurgitation. J Am Coll Cardiol. 2023 Feb 7;81(5):431-442. doi: 10.1016/j.jacc.2022.11.034. PMID 36725171
- [Derived] Lim DS, Smith RL, Gillam LD, Zahr F, Chadderdon S, Makkar R, von Bardeleben RS, Kipperman RM, Rassi AN, Szerlip M, Goldman S, Inglessis-Azuaje I, Yadav P, Lurz P, Davidson CJ, Mumtaz M, Gada H, Kar S, Kodali SK, Laham R, Hiesinger W, Fam NP, Kessler M, O'Neill WW, Whisenant B, Kliger C, Kapadia S, Rudolph V, Choo J, Hermiller J, Morse MA, Schofer N, Gafoor S, Latib A, Koulogiannis K, Marcoff L, Hausleiter J; CLASP IID Pivotal Trial Investigators. Randomized Comparison of Transcatheter Edge-to-Edge Repair for Degenerative Mitral Regurgitation in Prohibitive Surgical Risk Patients. JACC Cardiovasc Interv. 2022 Dec 26;15(24):2523-2536. doi: 10.1016/j.jcin.2022.09.005. Epub 2022 Sep 17. PMID 36121247